CLINICAL TRIAL: NCT00207636
Title: Community Interventions in Non-medical Settings to Increase Informed Decision Making for Prostate Cancer Screening - Harvard - SIP 21-04
Brief Title: Community Interventions in Non-medical Settings to Increase Informed Decision Making for Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDC-NCCDPHP-2504; NCT00137618 (obsolete NCT alias)
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: Computer-Assisted Decision Making; Workplace; Screening
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Distribution of printed materials
- Computer Assisted Decision making tool (Experimental): The intervention consisted of access to a computer tailored decision aid designed to promote informed decision making.
  Interventions: Behavioral: Computer Assisted Decision making tool

INTERVENTIONS:
Behavioral: Computer Assisted Decision making tool — The intervention consisted of access to a computer tailored decision aid designed to promote informed decision making.
  Arms: Computer Assisted Decision making tool

SUMMARY:
The purpose of this study is to develop and evaluate a computer-based decision aid (DA) for use by men considering prostate-specific antigen (PSA) screening for prostate cancer. Major medical organizations recommend that men discuss the risks and benefits of this test with their physician before making the decision. This educational, interactive DA will help them prepare for that discussion.

DETAILED DESCRIPTION:
Prostate cancer (CaP) is a formidable public health problem in the US and in industrialized countries worldwide. Methods for primary prevention of CaP are unknown. As a result, early detection has become a mainstay of cancer control efforts. However, there is considerable controversy regarding the efficacy of screening in reducing disease-specific mortality. In light of this uncertainty, major medical organizations, including the National Cancer Institute, currently recommend that men discuss the pros and cons of CaP screening and make individualized screening decisions with their health care providers. However, because of constraints on time during medical encounters, it is not always feasible for providers to engage in in-depth discussions regarding the complexities of this issue. Therefore, interventions to promote informed decision-making (IDM) outside of clinical settings are needed.

In this study, we propose to: (1) develop an interactive computer-based decision aid (DA) to promote IDM for CaP screening; and (2) conduct a randomized controlled worksite trial to evaluate the impact the DA intervention on employed men's ability to make informed decisions regarding CaP. This work is designed to be responsive to recent calls for IDM interventions in community settings among diverse populations. If successful, our findings could validate the effectiveness of DAs to promote IDM for CaP and serve as a model for widespread dissemination, thus improving quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Worksites employing at least 100 men in target age group (45-65 years old)

Exclusion Criteria:

* Worksites with high turnover
* Non-English speaking workers
* Temporary or contract workers

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2004-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Allen, PN MPH ScD, Principal Investigator — Dana-Farber Cancer Institute; Harvard School of Public Health
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Background] Allen JD, Othus MK, Hart A Jr, Tom L, Li Y, Berry D, Bowen D. A randomized trial of a computer-tailored decision aid to improve prostate cancer screening decisions: results from the Take the Wheel trial. Cancer Epidemiol Biomarkers Prev. 2010 Sep;19(9):2172-86. doi: 10.1158/1055-9965.EPI-09-0410. Epub 2010 Aug 17. PMID 20716619

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Distribution of printed material
- Experimental Group: The intervention is access to a computer-assisted decision-making tool designed to promote informed decision-making.
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 414 | 398
Completed | 334 | 291
Not Completed | 80 | 107

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: The intervention is access to a computer-assisted decision-making tool designed to promote informed decision-making.
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 414 | 398 | 812
Age, Customized [Count of Participants; unit: Participants]
  45 to 49 years old | 120 | 151 | 271
  50 to 54 years old | 126 | 106 | 232
  55 years old or older | 153 | 93 | 246
  Missing age | 15 | 48 | 63
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 414 | 398 | 812

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Were Ready to Make a Decision or Were Undecided
Description: Readiness to make a decision based on Stage of Decision-Making Scale (O'Connor A et al, 2008) with five responses ranging from "I haven't thought about it before" to "I have made a decision, and I am not likely to change my mind." Men were classified as having "decided" if they stated either that they had made a decision, but were willing to reconsider, or if they responded that they had made a decision but were unlikely to change their mind. Those "undecided" reported that they had not thought about the decision, or were uncertain.
Time Frame: Assessed at baseline and follow-up, up to 10 months
Measure: Count of Participants; unit: Participants
Groups:
- Control: Distribution of printed material
- Experimental: The intervention is access to a computer-assisted decision-making tool designed to promote informed decision-making.
Arm/Group | Control | Experimental
Number analyzed (Participants) | 334 | 291
Participants
  Decided : Baseline | 134 | 90
  Decided : Follow-up | 144 | 125
  Undecided : Baseline | 200 | 201
  Undecided : Follow-up | 190 | 166

2. Primary Outcome: Percentage of Correct Responses in Assessing Mens' Recognition of the Prostate-specific Antigen Test and Knowledge Related to Prostate-cancer Topics.
Description: Recognition of test based upon a standard single item and 14 validated questions assessed knowledge of prostate cancer prevalence, risk factors, screening modalities, diagnostic procedures, and treatment-related complications.
Time Frame: Assessed at baseline and follow-up, up to 10 months
Measure: Mean (Standard Error); unit: percentage of correct responses
Arm/Group | Control | Experimental
Number analyzed (Participants) | 334 | 291
percentage of correct responses
  Baseline | 56 (1.23) | 56 (2.68)
  Follow-up | 60 (1.6) | 66 (2.08)

3. Primary Outcome: Mean and Standard Error of a Scale Used to Assess Men's Confidence Level in Making Decisions Related to Prostate Cancer Screening.
Description: The confidence in ability to participate in decision making to the extent desired using the 11-item Decision Self-Efficacy Scale was assessed. Respondents were asked to reflect on their confidence level about various aspects of the decision-making process, with response options of "very confident" (score = 4) to "not at all confident" (score = 0). Scores were summed, divided by 11, and multiplied by 25, to arrive at a range of scores from 0 (no self-efficacy) to 100 (higher self-efficacy).
Time Frame: Assessed at baseline and follow-up, up to 10 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 334 | 291
score on a scale
  Baseline | 79 (1.59) | 83 (2.46)
  Follow-up | 79 (1.81) | 83 (2.36)

4. Primary Outcome: Percentage of Consistency Between Screening Preference and Personal Values Relevant to the Screening Decision
Description: Items were developed to assess the personal importance or relative worth of the advantages and limitations of screening based on focus group themes and published literature. Some to the themes include: importance of information, accuracy of test, potential side effects of treatment.
Time Frame: Assessed at baseline and follow-up, up to 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 334 | 291
Participants
  Consistent: Baseline | 244 | 207
  Consistent: Follow-up | 247 | 201
  Inconsistent : Baseline | 87 | 81
  Inconsistent : Follow-up | 80 | 90
  Missing: Baseline | 3 | 3
  Missing: Follow-up | 7 | 1

5. Secondary Outcome: Percentage of Men Who Have Active Decision-making, Collaborative Decision-making, or Passive Decision-making Styles
Description: Assessed through the Control Preferences Scale (Degner LF et al, 1997). Individuals were assessed who should make medical decisions. The active decision-making category included responses where men made the final decision on their own or after considering their doctor's opinions. The collaborative decision-making category included responses where men and their doctors shared the responsibility for the decision. The passive decision-making category included responses where the doctors made the final decision after considering a man's input or that the doctor made the final decision.
Time Frame: Assessed at baseline and follow-up, up to 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 334 | 291
Participants
  Baseline: active/collaborative | 305 | 274
  Follow-up: active/collaborative | 308 | 277
  Baseline: passive | 28 | 15
  Follow-up: passive | 23 | 13
  Baseline: missing | 1 | 2
  Follow-up: missing | 3 | 1

6. Secondary Outcome: Mean and Standard Error of a Scale to Measure Decisional Conflict
Description: Measured through the Decisional Conflict Scale (O'Connor AM et al, 2003) by rating statements related to decision making and responding on a five-point scale ranging from "strongly agree' to "strongly disagree". Scales were standardized from 0 (no conflict) to 100 (extreme conflict).
Time Frame: Assessed at baseline and follow-up, up to 10 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 334 | 291
score on a scale
  Baseline | 28 (2.12) | 25 (2.08)
  Follow-up | 20 (2.07) | 14 (2.01)

ADVERSE EVENTS:
Time Frame: This was an intervention trial, so no adverse events were not monitored or assessed.
Description: This was an intervention trial, so no adverse events were not monitored or assessed.
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. Overall use of the decision aid in the intervention group was lower.
2. Findings may not be generalizable to since study population was predominantly white and employed.
3. A new scale for decisional consistency was used.
4. Self-report values of prostate-specific antigen testing were used.
5. Short-term changes (3-months) were measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No